CLINICAL TRIAL: NCT00770822
Title: A Multicenter Clinical Study of the Sonablate® 500 (SB-500) for the Treatment of Localized (T1c/T2a) Prostate Cancer With HIFU
Brief Title: Clinical Study of the Sonablate® 500 to Treat Localized (T1c/T2a) Prostate Cancer
Acronym: SetPace
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SonaCare Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSI-002; NCT00485381 (obsolete NCT alias)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
Keywords: Primary; Prostate; Cancer; Primary T1c/T2a organ confined prostate cancer; organ-confined
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device, HIFU (Experimental): High Intensity Focused Ultrasound
  Interventions: Device: HIFU (Sonablate® 500)
- Device, brachytherapy (Active Comparator): Brachytherapy
  Interventions: Device: Brachytherapy

INTERVENTIONS:
Device: HIFU (Sonablate® 500) — High Intensity Focused Ultrasound
  Other Names: SB-500; Sonablate 500; HIFU
  Arms: Device, HIFU
Device: Brachytherapy — Standard of care
  Other Names: Raditation Seed Implants; Brachy
  Arms: Device, brachytherapy

SUMMARY:
This study will compare high intensity focused ultrasound to standard brachytherapy in the treatment of primary, organ confined prostate cancer.

DETAILED DESCRIPTION:
The proposed study is a prospective, non-randomized concurrently controlled study. The active treatment arm uses the HIFU procedure with the Sonablate device. The control arm uses the brachytherapy procedure. The safety and effectiveness of the Sonablate arm will be compared with the brachytherapy arm. The control arm of the study will be conducted at clinical sites different from the Sonablate arm.

ELIGIBILITY:
Inclusion Criteria:

* T1c or T2a carcinoma of the prostate confirmed by biopsy;
* life expectancy of 5(five) years or more;
* prostate biopsy with 10(ten) or more core biopsies;
* Gleason score of 6(six) or less;
* serum Prostate Specific Antigen (PSA) of 10(ten)ng/ml or less;
* prostate volume of less than 40(Forty)cc;
* distance from the Anterior capsule surface to the Posterior capsule surface (AP Diameter) of 40(Forty)cm or less;
* informed consent for the treatment study through 24 months post-treatment follow-up

Exclusion Criteria:

* men who have had previous definitive treatment for prostate cancer;
* evidence of metastatic disease and/or a previous positive bone-scan, previous diagnosis or treatment for cancer within the last 5(five) years;
* prior hormonal therapy for prostate cancer (including bilateral orchiectomy);
* inability to tolerate a transrectal ultrasound;
* active urinary tract infection;
* functional bladder problems;
* prior significant rectal surgery;
* intra-prostatic calcifications greater than 1(One)cm in diameter;
* interest in future fertility;
* prostatic surgery/procedure (except biopsy) within 1(One) year;
* large median lobe of the prostate;
* use of medications that can affect PSA within 2(Two) months (e.g. finasteride, saw palmetto);
* current bladder cancer, urethral stricture, or bladder neck contracture;
* urinary tract and/or rectal fistula;
* rectal fibrosis/stenosis;
* anomaly of the rectal anatomy or mucus membrane;
* prostate seroma/abcess;
* prostatitis;
* compromised renal function or upper urinary tract disease secondary to urinary obstruction;
* bleeding disorders/coagulopathy based on measures of PT and PTT;
* implant in the prostate or within 1(One)cm of the prostate;
* zip code of the primary residence of the subject is greater than 200(Two hundred) miles from the clinical site or transportation that would hinder the completion of the study

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2007-04; Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the absence of biochemical failure, which is defined as a rise of 2.0 ng/mL or more above the PSA nadir and negative biopsy at 24 months. | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schoenberg, M.D., Principal Investigator — Johns Hopkins Medical Institution
Locations (6):
- United States (6):
  - Brachytherapy Site: Urology Centers of Alabama, Birmingham, Alabama
  - Brachytherapy Site: Specialists in Urology, Naples, Florida
  - Brachytherapy Site: Grand Strand Urology, Myrtle Beach, South Carolina
  - HIFU Site: Southeast Urology Network, Memphis, Tennessee
  - HIFU Site: Urology Associates, Nashville, Tennessee
  - HIFU Site: Urology of San Antonio, San Antonio, Texas